CLINICAL TRIAL: NCT02800941
Title: Bleeding Frequency Under Anticoagulant Treatment in Pulmonary Hypertension : HEMA-HTP Multicentric Study.
Brief Title: Bleeding Frequency Under Anticoagulant Treatment in Pulmonary Hypertension
Acronym: HEMA-HTP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1608037; 2016-001608-41 (EudraCT Number)
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial hypertension; Oral anticoagulants; Major bleedings
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Warfarin; fluindione; Acenocoumarol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oral anticoagulant treatment: Patients with pulmonary hypertension are treated with oral anticoagulants according to the usual practice. Patients have follow-up at 3, 6 and 12 months.
  Interventions: Drug: Oral anticoagulant treatment

INTERVENTIONS:
Drug: Oral anticoagulant treatment — The treatment is delivered according to the usual practice.
  Other Names: warfarin (Coumadine®); fluindione (Préviscan®); acenocoumarol (Sintrom®)

SUMMARY:
Pulmonary hypertension (PHT) patients often receive long term oral anticoagulants. If the indication is strong, in the secondary chronic thrombo-embolism pulmonary hypertension (CTE-PHT) prevention, the frequent prescription (50 to 90% of patients) contrasts with their low level of proof in the PHT. Last but not least, anticoagulants are known to be the principal cause of iatrogenic hospitalization (major bleeding).

In this study, patients are all followed during one year, to determine the annual frequency of major bleedings (according to the International Society on Thrombosis and Haemostasis (ISTH) international definition). Each event notified is validated by an independent committee for clinical events.

DETAILED DESCRIPTION:
Pulmonary hypertension (PHT) patients often receive long term oral anticoagulants. If the indication is strong, in the secondary chronic thrombo-embolism pulmonary hypertension (CTE-PHT) prevention, the frequent prescription (50 to 90% of patients) contrasts with their low level of proof in the PHT. Last but not least, anticoagulants are known to be the principal cause of iatrogenic hospitalization (bleeding).

The only one study scaling the tolerance of anticoagulants for this population found major hemorrhagic levels discording with the clinical practice : really high for connectives associated to pulmonary arterial hypertension (PAHT), and lower in "simple" pulmonary embolism in CTE-PHT. These discoveries could belong to methodological failures of this study: a retrospective, monocentric one, without adjudication of events by an independent committee. Furthermore, there were no information about the existence of a validated indication for anticoagulant treatments.

Patients are all followed during one year, to determine the annual frequency of major bleedings (according to the International Society on Thrombosis and Haemostasis (ISTH) international definition). Each event notified is validated by an independent committee for clinical events.

ELIGIBILITY:
Inclusion Criteria:

* Patient insured or entitled to a social security scheme;
* Patient with confirmed pulmonary hypertension;
* Pulmonary hypertension among the following etiological diagnosis: idiopathic PAH, PAH associated with appetite suppressants, PAH associated with connective, or Chronic Thrombo-embolism Pulmonary Hypertension;
* Patients receiving oral anticoagulants.

Exclusion Criteria:

* Impossible following;
* Bleeding at baseline;
* Life expectancy of less than 3 months;
* Pulmonary hypertension in Group 2, Group 3 (in the absence of associated pulmonary embolism) and Group 5 (in the absence of associated pulmonary embolism).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of pulmonary hypertension patients receiving oral anticoagulant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Number of major bleeding (according to the International Society on Thrombosis and Haemostasis definition) | 1 year
  Major bleedings (according to the International Society on Thrombosis and Haemostasis definition) will be notified during one year under oral anticoagulant treatment.

SECONDARY OUTCOMES:
Number of clinically relevant bleedings | 1 year
  Clinically relevant bleedings (major and non major ones) will be notified during one year under oral anticoagulant treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bertoletti, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (4):
- France (4):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Grenoble, Grenoble
  - Hospices Civils de Lyon, Lyon
  - CHU de Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No